CLINICAL TRIAL: NCT01604122
Title: Cross-sectional, Non-interventional Burden Of Disease (Bod) Study In Patients With Transthyretin Familial Amyloidosis Polyneuropathy (Ttr-fap) Or Transthyretin Cardiomyopathy (ttr-cm) And Caregivers
Brief Title: Burden of Disease Study In Patients With Transthyretin Familial Amyloidosis Polyneuropathy (TTR-FAP) orTransthyretin Cardiomyopathy (TTR-CM) And Caregivers
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461036
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2017-03

CONDITIONS: Transthyretin Familial Amyloidosis Polyneuropathy (TTR-FAP); Transthyretin Cardiomyopathy (TTR-CM); Familial Amyloid Cardiomyopathy; Senile Systemic Amyloidosis (SSA)
Keywords: Survey; burden of illness; caregivers; TTR-FAP; TTR-CM; familial amyloid polyneuropathy; observational; transthyretin familial amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with TTR-FAP or TTR-CM. No drug will be administered; this is a non-interventional observational study.
  Interventions: Other: No drug
- Caregivers: Caregivers who are taking care of patients with TTR-FAP or TTR-CM. No drug will be administered; this is a non-interventional observational study.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — No drug.
  Groups: Patients
Other: No drug — No drug.
  Groups: Caregivers

SUMMARY:
This study is an online (web-based) or paper-based survey for patients with transthyretin familial amyloidosis polyneuropathy (TTR-FAP) and caregivers. The results will be used to describe the emotional, physical, and financial impact of having TTR-FAP or caring for someone who has the disease.

DETAILED DESCRIPTION:
Convenience sample of patients and caregivers recruited through patient advocacy groups. Convenience sample.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18-85 years inclusive) diagnosed with TTR-FAP or TTR-CM and experiencing symptoms or currently providing care for a patient with TTR-FAP or TTR-FAP

Exclusion Criteria:

* Caregivers who formally care for a TTR-FAP or TTR-CM patient as part of their job description and receive payment for their services.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (ages 18-85 years inclusive) diagnosed with TTR-FAP or TTR-CM and experiencing symptoms or currently providing care for a patient with TTR-FAP or TTR-CM
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-04-18 (Actual); Primary Completion 2015-07-27 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Stewart M, Shaffer S, Murphy B, Loftus J, Alvir J, Cicchetti M, Lenderking WR. Characterizing the High Disease Burden of Transthyretin Amyloidosis for Patients and Caregivers. Neurol Ther. 2018 Dec;7(2):349-364. doi: 10.1007/s40120-018-0106-z. Epub 2018 Aug 2. PMID 30073497

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Diagnosed With ATTR: Participants diagnosed with transthyretin amyloidosis (ATTR) with two phenotypes: familial amyloid polyneuropathy (TTR-FAP) and cardiac amyloidosis (TTR-CM) were included in this non-interventional study to complete the one time survey.
- Caregivers: Caregivers were those participants who provided support and care to the participants diagnosed with ATTR (TTR-FAP and TTR-CM) and completed the caregiver survey, regardless of whether they themselves were diagnosed with ATTR or not.
Period: Overall Study
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Started | 60 | 32
Completed | 60 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study and completed the survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Diagnosed With ATTR | Caregivers | Total
Number analyzed (Participants) | 60 | 32 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.0) | 55.9 (12.8) | 57.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 22 | 35
  Male | 47 | 10 | 57

OUTCOME MEASURES:

1. Primary Outcome: Demographical Characteristics of Participants
Description: Main characteristics included were education level and employment status which were asked from all participants and caregivers. Type of job (full-time, part-time) was asked only from those participants and caregivers who provided their employment status as employed. Those who were unemployed reported their cause of unemployment, whether it was due to ATTR or not.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'n' signifies those participants who were evaluable for specific category for each arm respectively.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 60 | 32
participants
  Employment Status: Currently Employed (n= 60, 32) | 20 | 11
  Employment Status:Not Currently Employed (n=60,32) | 39 | 19
  Employment Status: Skipped (n= 60, 32) | 1 | 1
  Employment Status: Not Asked (n= 60, 32) | 0 | 1
  Employment Type: Full-Time (n= 20, 11) | 11 | 9
  Employment Type: Part-Time (n= 20, 11) | 9 | 2
  Unemployed: Due to ATTR (n= 39, 19) | 25 | 0
  Unemployed: Not due to ATTR (n= 39, 19) | 13 | 0
  Unemployed: Skipped (n= 39, 19) | 1 | 0
  Unemployed: Not Asked (n= 39, 19) | 0 | 19
  Education Level: Lower Than High School (n=60,32) | 6 | 3
  Education Level: High School/Equivalent(n=60,32) | 8 | 6
  Education Level: Associate Degree(n=60,32) | 12 | 3
  Education Level: College Degree (n= 60, 32) | 14 | 10
  Education Level: Professional or Graduate(n=60,32) | 20 | 7
  Education Level: Skipped (n= 60, 32) | 0 | 2
  Education Level: Not Asked (n= 60, 32) | 0 | 1

2. Primary Outcome: Disease Characteristics of Participants: Disease Duration
Description: Duration of disease was defined as the time from diagnosis of disease until baseline visit. This outcome measure was planned to be assessed for reporting arm of participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey.
Measure: Median (Full Range); unit: years
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
years | 5.6 (4.0) [0.0 to 16.1]

3. Primary Outcome: Disease Characteristics of Participants: Mutation Type
Description: Genetic mutation leads to misfolding of protein transthyretin (TTR) which results in ATTR. In this outcome, number of participants with each type of resulted mutation type (Val30Met, wild type TTR, Phe64Leu, Ser77Tyr, Thr60Ala or other than these) were reported. This outcome was planned to be assessed for reporting arm of participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
participants
  Val30Met | 18
  Wild Type TTR | 2
  Phe64Leu | 4
  Ser77Tyr | 3
  Thr60Ala | 11
  Other | 5
  Unknown | 17

4. Primary Outcome: Disease Characteristics of Participants: Liver Transplantation Status
Description: TTR protein is primarily synthesized in the liver. Liver transplantation was considered as one of the measure to eliminate the main source of variant TTR. In the study, participants who were diagnosed with ATTR were asked for their liver transplantation status (whether they had transplantation or not). In this outcome measure, number of participants with liver transplant status were reported. This outcome was planned to be assessed for reporting arm of participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
participants
  With Liver Transplantation | 31
  No Liver Transplantation | 29

5. Primary Outcome: Disease Characteristics of Participants: Number of Participants With Family History of ATTR
Description: Family history of participants diagnosed with ATTR was assessed to determine whether family history of ATTR was a significant risk factor for ATTR or not. This outcome was planned to be assessed for reporting arm of participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
participants | 51

6. Primary Outcome: Disease Characteristics of Participants: Mobility Status
Description: Mobility, i.e., ability to walk was assessed as a part of loss of functioning in the participants diagnosed with ATTR. In this outcome, number of participants with their different mobility status along with the use of mobility aids (able to walk normally, some problems with feet but able to walk without difficulty, some difficulty walking but can walk without help, confined to bed all the time, need 1 cane or crutch to walk, need 2 canes/crutches or a walker to walk) were reported.
Time Frame: Baseline (Day 1)
Population: All participants who were included in the study and completed the survey.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
participants
  Able to Walk Normally | 15
  Some Problems: Able to Walk Without Difficulty | 16
  Some Difficulty: Can Walk Without Help | 14
  Need 1 Cane or Crutch to Walk | 6
  Need 2 Canes/Crutches or a Walker to Walk | 9
  Confined to bed all the Time | 0

7. Primary Outcome: 12-Item Short-Form Health Survey (SF-12) Scores
Description: SF-12 was a patient reported outcome survey that represented overall health status by measuring 8 health-related aspects of an individual: Body pain, general mental health, perception of general health, physical functioning, role limitations caused by mental condition, role limitations caused by a physical condition, social functioning, and vitality. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. Responses on the SF-12 were also used to calculate 2 summary scores: Physical component score (PCS) and mental component score (MCS). The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health), where 100 indicated good health condition.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'n' signifies those participants who were evaluable for specific component for each arm respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 60 | 32
units on a scale
  Physical Health Summary (n= 56, 28) | 33.6 (11.5) | 42.2 (13.7)
  Mental Health Summary (n= 56, 28) | 47.1 (10.8) | 39.3 (11.1)
  Physical Functioning (n= 58, 29) | 32.2 (11.0) | 43.1 (13.7)
  Role-Physical (n= 56, 28) | 33.7 (10.7) | 39.1 (13.1)
  Bodily Pain (n= 57, 29) | 43.0 (13.3) | 39.5 (15.3)
  General Health (n= 59, 29) | 37.2 (12.0) | 39.8 (13.5)
  Vitality (n= 56, 29) | 41.1 (10.6) | 45.7 (11.5)
  Social Functioning (n= 57, 29) | 41.0 (11.6) | 39.5 (13.8)
  Role-Emotional (n= 57, 29) | 39.5 (13.9) | 34.3 (13.6)
  Mental Health (n= 57, 29) | 48.2 (10.2) | 41.8 (11.4)

8. Primary Outcome: Hospital Anxiety and Depression Scale (HADS): Depression and Anxiety Subscale Scores
Description: HADS: participant rated 14-item questionnaire with 2 subscales; HADS-anxiety scale (HADS-A) and HADS-depression scale (HADS-D). HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items and the participant responds as to how each item applies to him/her over the past week prior to baseline visit, on 4-point response scale. Separate scores were calculated for anxiety and depression with score ranges from 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score range was from 0 to 21 for each subscale; higher score indicating greater severity of anxiety and depression symptoms.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 55 | 29
units on a scale
  Depression Sub-Scale | 5.9 (3.4) | 8.1 (5.3)
  Anxiety Sub-Scale | 5.9 (3.9) | 10.8 (4.5)

9. Primary Outcome: Euro Quality of Life (EQ-5D-3L)- Health State Profile Utility Score
Description: EQ-5D-3L: participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. For utility score, participants rated their current health state on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with each dimension having three levels of function: 1 indicates no problem; 2 indicates some problem; 3 indicates extreme problem. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total score range of 0.05 to 1.00; higher scores indicating a better health state.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'N' signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 57 | 28
units on a scale | 0.74 (0.20) | 0.65 (0.33)

10. Primary Outcome: Euro Quality of Life (EQ-5D-3L)- Visual Analog Scale (VAS) Score
Description: EQ-5D: participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. The VAS component rated the current health state on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicating a better health state.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 55 | 28
units on a scale | 58.7 (19.8) | 64.2 (28.1)

11. Primary Outcome: Work Productivity and Activity Impairment- Specific Health Version (WPAI-SH): Percent of Work Time Missed
Description: The WPAI assesses work productivity and impairment. It was a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days prior to baseline visit. The questionnaire asked about current employment status, hours worked, hours missed from work and degree to which a specified health problem (ATTR) or caregiving affected work productivity and regular activities. Percentage of work time missed of participants were recorded and reported.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Median (Full Range); unit: percentage of work time missed
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 18 | 9
percentage of work time missed | 2 (26.0) [0 to 79] | 0 (21.8) [0 to 57]

12. Primary Outcome: Work Productivity and Activity Impairment- Specific Health Version: Percent Impairment While Working
Description: The WPAI assesses work productivity and impairment. It was a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days prior to baseline visit. The questionnaire asks about current employment status, hours worked, hours missed from work and degree to which a specified health problem (ATTR) or caregiving affected work productivity and regular activities. Component scores included percent work time missed due to the health problem; percent impairment while working due to problem; percent overall work impairment due to problem; and percent activity impairment due to problem. The computed percentage range for each sub-scale was from 0-100, where higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 18 | 8
units on a scale | 32.8 (32.7) | 36.3 (31.6)

13. Primary Outcome: Work Productivity and Activity Impairment- Specific Health Version: Percent Overall Work Impairment
Description: The WPAI assesses work productivity and impairment. It was a 6-item questionnaire used to assess the degree to which a specified health problem affected work productivity and regular activities over the past 7 days prior to baseline visit. The questionnaire asked about current employment status, hours worked, hours missed from work and degree to which a specified health problem (ATTR) or caregiving affected work productivity and regular activities. Component scores included percent work time missed due to the health problem; percent impairment while working due to problem; percent overall work impairment due to problem; and percent activity impairment due to problem. The computed percentage range for each sub-scale was from 0-100, where higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 18 | 8
units on a scale | 37.3 (36.1) | 40.4 (35.6)

14. Primary Outcome: Work Productivity and Activity Impairment- Specific Health Version: Percent Activity Impairment
Description: as for outcome 12
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 55 | 17
units on a scale | 49.8 (30.5) | 41.2 (30.4)

15. Primary Outcome: Healthcare Resource Use Survey: Number of Outpatient Visits to Healthcare Providers
Description: Healthcare resources use survey of participants diagnosed with ATTR and caregivers was assessed by questions concerning a variety of different types of treatment and resources including outpatient visits to healthcare providers, hospitalizations, emergency/urgent care visits, symptomatic treatments, and out-of-pocket costs (for example, costs of travel to receive care).
Time Frame: Baseline (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: outpatient visits
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 60 | 32
outpatient visits
  Primary Care Provider/Family Doctor (n=27, 12) | 2.0 (1.5) | 1.8 (1.5)
  Neurologist (n=12, 6) | 1.4 (0.8) | 1.2 (0.4)
  Cardiologist (n=17, 9) | 2.2 (2.7) | 1.1 (0.3)
  Gastroenterologist (n=9, 3) | 1.3 (0.5) | 1.3 (0.6)
  Hematologist (n=5, 4) | 2.8 (0.8) | 1.8 (1.5)
  Liver Transplant Surgeon (n=6, 5) | 1.2 (0.4) | 1.0 (0.0)
  Nurse/Nurse Practitioner (n=9, 5) | 4.4 (5.6) | 2.6 (2.2)
  Urologist (n=9, 1) | 1.9 (1.3) | 2.0 (NA) — Data for standard deviation was not estimable as only 1 participant was analyzed for this measure.
  Ophthalmology (n=5, 1) | 1.0 (0.0) | 2.0 (NA) — Data for standard deviation was not estimable as only 1 participant was analyzed for this measure.
  Other (n=18, 6) | 2.2 (2.8) | 1.0 (0.0)

16. Primary Outcome: Healthcare Resource Use Survey: Number of Hospitalizations
Description: as for outcome 15
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hospitalization visits
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 9 | 6
hospitalization visits | 2.1 (2.0) | 3.5 (1.9)

17. Primary Outcome: Healthcare Resource Use Survey: Number of Emergency Care Visits
Description: as for outcome 15
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: emergency care visits
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Number analyzed (Participants) | 13 | 6
emergency care visits | 1.3 (0.9) | 2.8 (1.3)

18. Primary Outcome: Healthcare and Resource Use Survey: Symptomatic Treatment of Participants
Description: Healthcare resources use survey of participants diagnosed with ATTR was assessed by questions concerning a variety of treatments and resources included outpatient visits to healthcare providers, hospitalizations, emergency/urgent care visits, symptomatic treatments, and out-of-pocket costs. Number of participants (diagnosed with ATTR) who visited non-medical practitioners (nutrition consultant/dietician, chiropractor, acupuncturist, massage therapist, occupational therapist or other than these) for symptomatic treatments were reported.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey.
Measure: Number; unit: participants
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
participants | 12

19. Primary Outcome: Healthcare Resource Use Survey: Number of Symptomatic Treatment Visits
Description: Healthcare resources use survey of participants diagnosed with ATTR was assessed by questions concerning a variety of treatments and resources included outpatient visits to healthcare providers, hospitalizations, emergency/urgent care visits, symptomatic treatments, and out-of-pocket costs. Number of visits of participants (diagnosed with ATTR) who visited non-medical practitioners (nutrition consultant/dietician, chiropractor, acupuncturist, massage therapist, occupational therapist or other than these) for symptomatic treatments were reported.
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'N' signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for specific category.
Measure: Mean (Standard Deviation); unit: symptomatic treatment visits
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 12
symptomatic treatment visits
  Nutrition Consultant/Dietitian (n=2) | 4.0 (2.8) [2 to 6]
  Chiropractor (n=1) | 1.0 (NA) [1 to 1] — Data for standard deviation was not estimable as only 1 participant was analyzed for this measure.
  Acupuncturist (n=3) | 3.7 (2.5) [1 to 6]
  Massage Therapist (n=5) | 3.0 (1.9) [1 to 6]
  Occupational Therapist (n=2) | 3.5 (3.5) [1 to 6]
  Other (n=3) | 2.0 (1.0) [1 to 3]

20. Primary Outcome: Healthcare Resource Use Survey: Out-of-Pocket Costs
Description: Healthcare resources use survey of participants diagnosed with ATTR was assessed by questions concerning a variety of treatments and resources included outpatient visits to healthcare providers, hospitalizations, emergency/urgent care visits, symptomatic treatments, and out-of-pocket costs (expenditure on nutritional supplements, non-prescription medications and travel to receive medical care).
Time Frame: Baseline (Day 1)
Population: All participants who were enrolled in the study and completed the survey. Here, 'n' signifies those participants who were evaluable for specific category.
Measure: Median (Full Range); unit: dollars
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 60
dollars
  Nutritional Supplements (n=13) | 150 (121) [30 to 450]
  Non-Prescription Medications (n=46) | 28 (76) [0 to 300]
  Travel to Receive Medical Care (n=45) | 30 (823) [0 to 4000]

21. Primary Outcome: Participants Pain Score
Description: Participants diagnosed with ATTR rated their pain due to the health condition based on 3 items: pain right now, average pain in the past week, and worst pain in the past week prior to baseline visit. All 3 items were rated on an 11-point numeric rating scale ranging from 0=none to 10=severe pain, where higher scores indicated severe pain.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 39
units on a scale
  Pain Right now | 3.1 (3.1)
  Average Pain Past Week | 3.4 (3.0)
  Worst Pain Past Week | 4.3 (3.4)

22. Primary Outcome: Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QOL-DN) Total Quality of Life (TQOL): Total Scores
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire used to assess impact of neuropathy on the quality of life of participants diagnosed with ATTR. Scoring was based on 35 questions that yield a TQOL as well as 5 subscale scores: activities of daily living, large fiber neuropathy/physical functioning, small fiber neuropathy, autonomic neuropathy, and symptoms. TQOL= sum of all the items, total possible score range= -2 to 138, where higher score=worse quality of life. This outcome measure was planned to be analyzed only for the reporting arm of participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 47
units on a scale | 54.6 (32.8)

23. Primary Outcome: Norfolk Quality of Life-Diabetic Neuropathy Total Quality of Life: Subscale Scores
Description: Norfolk QOL-DN: 35-item participant-rated questionnaire used to assess impact of neuropathy on the quality of life of participants diagnosed with ATTR. It was summarized in 5 domains: (1) Activities of daily living (score ranges from 0 to 20, where higher score=worse quality of life); (2) Large fiber neuropathy/physical functioning (score ranges from -2 to 58, where higher score=worse condition); (3) Small fiber neuropathy (score ranges from 0 to 16, where higher score=worse condition); (4) Autonomic neuropathy (score ranges from 0 to 12, where higher score=worse condition) and (5) Symptoms (score ranges from 0 to 32, where higher score=less symptoms of disease). Total possible score range= -2 to 138, where higher score=worse quality of life. This outcome measure was analyzed only for the participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 54
units on a scale
  Symptoms (n= 50) | 11.5 (7.4)
  Activities of Daily Living (n= 50) | 5.7 (6.1)
  Small Fiber Neuropathy (n= 49) | 6.0 (4.2)
  Large Fiber Neuropathy (n= 47) | 26.5 (16.8)
  Autonomic Neuropathy (n= 50) | 4.2 (3.1)

24. Primary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ) Scores
Description: KCCQ was a 23-item participant-completed questionnaire that assessed health status and health-related quality of life (HRQoL) in participants with heart failure. It was quantified in to following 10 summary scores: physical limitation, symptom frequency, symptom severity, and symptom stability, total symptoms, quality of life, social interference, self-efficacy, overall summary and clinical summary. Each summary score was scaled to range from 0 (minimum) to 100 (maximum), with higher scores representing greater disability. Total score ranged from 0 to 100, where higher scores indicated better functioning, fewer symptoms, and better disease specific quality of life.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Diagnosed With ATTR
Number analyzed (Participants) | 17
units on a scale
  Physical Limitation Score | 41.7 (29.2)
  Symptom Stability Score | 48.5 (10.7)
  Symptom Frequency Score | 47.7 (25.1)
  Symptom Burden Score | 51.0 (24.5)
  Total Symptom Score | 49.3 (23.8)
  Self-Efficacy Score | 78.7 (21.1)
  Quality of Life Score | 50.0 (18.6)
  Social Limitation Score | 31.8 (25.0)
  Overall Summary Score | 43.2 (20.0)
  Clinical Summary Score | 45.5 (25.2)

25. Primary Outcome: Zarit Burden Interview (ZBI): Total Scores
Description: ZBI was a 22-item questionnaire designed to evaluate five broad aspects of caregiver burden in terms of personal and role strain associated with caregiving. Five broad aspects were: burden in the relationship, emotional well-being, social and family life, finances, loss of control over one's life. Each item rated on a 5 point scale anchored at 0 for "never" and 4 for "nearly always." Total score ranges from 0-88 with higher scores indicating increased burden of care.
Time Frame: Baseline (Day 1)
Population: All participants who were included in the study and completed the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 32
units on a scale | 28.8 (17.5)

26. Primary Outcome: Zarit Burden Interview: Subscale Scores
Description: A questionnaire designed to evaluate aspects of caregiver burden in terms of personal and role strain associated with caregiving. Total score of ZBI scale ranges from 0-88 with higher scores indicating increased burden of care. Five subscale scores were also calculated: (1) Burden in the relationship (consist of 6-items, ranging from 0 to 24 where higher scores indicating increased burden in relationship); (2) Emotional well-being (consisting of 7-items, ranging from 0 to 28 where higher scores indicating worse condition; (3) Social and family life (consisting of 4-items, ranging from 0 to 16 where higher scores indicating worse life condition); (4) Finances (consisting of a single item, scored from 0 to 4 where higher scores indicating worse financial condition); and (5) Loss of control over one's life (consisting of 4-items, ranging from 0 to 16 where higher scores indicating worse control over life).
Time Frame: Baseline (Day 1)
Population: All participants who were included in the study and completed the survey. Here, 'n' signifies those participants who were evaluable for specific category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregivers
Number analyzed (Participants) | 32
units on a scale
  Burden in Relationship (n=28) | 7.6 (5.0)
  Emotional Well-Being (n=29) | 8.3 (5.9)
  Social and Family Life (n=28) | 5.1 (3.4)
  Finances (n=29) | 1.9 (1.4)
  Loss of Control Over Life (n=29) | 6.5 (3.5)

27. Primary Outcome: Caregiver Burden Items Assessment: Number of Hours Per Week Spent in Care of the Participants With ATTR
Description: Caregivers completed a series of questions related to the number of hours per week spent on providing care and support to the participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours per week
Arm/Group | Caregivers
Number analyzed (Participants) | 29
hours per week | 72 [2 to 168]

28. Primary Outcome: Caregiver Burden Items Assessment: Work Time Lost
Description: Caregivers completed a series of questions related to the loss in their working time while providing care and support to the participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Caregivers
Number analyzed (Participants) | 26
hours | 22 [0 to 168]

29. Primary Outcome: Caregiver Burden Items Assessment: Total Cost
Description: Caregivers completed a series of questions related to the total cost spent on providing healthcare support to participants diagnosed with ATTR.
Time Frame: Baseline (Day 1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Caregivers
Number analyzed (Participants) | 20
dollars | 9313.0 (33226.1) [0 to 150000]

ADVERSE EVENTS:
Description: Due to the non-interventional nature of the study, adverse events were not collected during the study.
Arm/Group | Participants Diagnosed With ATTR | Caregivers
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.